CLINICAL TRIAL: NCT01939041
Title: Efficacy of Unilateral Versus Bilateral Approach to Robot-Assisted Rehabilitation on Motor Control/Performance, Daily Functions, and Physiological Responses in Patients With Subacute Stroke
Brief Title: Efficacy of Unilateral Versus Bilateral Approach to Robot-Assisted Rehabilitation in Patients With Subacute Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult to recruit participant
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101-5194A3
Record Dates: First submitted 2013-08-21; First posted 2013-09-11 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2016-06

CONDITIONS: Subacute Stroke
Keywords: Subacute Stroke; Unilateral Robot-Assisted Training; Bilateral Robot-Assisted Training; Motor control; Physiological Response

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Robot-assisted therapy with InMotion3 (IMT) (Experimental): We will use the InMotion3 Wrist Robot (Figure 1) for the IMT group. During the InMotion3 therapy (IMT) session, participants will receive 5-minute of muscle tone normalization preparation and passive range of motion, then a 70-minute robot-assisted training followed by a 15-minute functional training. During the robot-assisted training, only the paretic hand will be trained and the participant will rest the forearm and hand on a cradle and the wrist and hand in a fixed positions. During the practice, a visual display will provide online visual feedback of accuracy and coordination success. And summary scores regarding movement accuracy and movement smoothness will be shown on the display periodically. After each IMT session, a 15 min functional task practice will be provided as described in the previous paragraph.
  Interventions: Device: InMotion3 (IMT)
- Robot-assisted therapy with Bi-Manu-Track (BMT) (Experimental): During the Bi-Manu-Track training (BMT), participant will use both nonparetic and paretic hands. Participants will receive 5-munite of muscle tone normalization preparation and passive range of motion, then will practice about 5-minute in Mode 1, 25-minute in Mode 2, and 5-minute in Mode 3 in wrist and forearm respectively. The training repetitions of each mode fall within the range of the protocols used in previous studies which would not cause adverse events (Hesse et al., 2005). The total minutes of each robot-assisted will be 70 minutes. After each BMT session, a 15 min functional task practice will be provided based on the same principles as the one in the IMT group.
  Interventions: Device: Bi-Manu-Track (BMT)
- Control intervention group (CI) (Active Comparator): The control group's therapy will be designed to control for the duration and intensity of the robot-assisted training (90 min/day, 5 days/wk, for 4 wk). The therapeutic activities in the control group will involve passive range of motion, weight bearing, stretching, strengthening of the paretic arm, gross motor activities, coordination tasks, unilateral and bilateral fine motor tasks, transition, mobility, and posture/balance.
  Interventions: Behavioral: Control intervention (CI)

INTERVENTIONS:
Device: InMotion3 (IMT) — Participant will practice about 2-5-minute of passive, 25-30-minute of assisted-active, and 3-5-minute of active motions in wrist and forearm respectively. The wrist motions will include flexion, extension, radial deviation, and ulnar deviation. Forearm motions will include supination and pronation. During the practice, a visual display will provide online visual feedback of accuracy and coordination success.
  Other Names: InMotion3 Wrist Robot; INMOTION Mechanical chair; INTERACTIVE MOTION TECHNOLOGIES, INC
  Arms: Robot-assisted therapy with InMotion3 (IMT)
Device: Bi-Manu-Track (BMT) — The Bi-Manu-Track enables the symmetrical practice of 2 movement patterns in conjunction with computer games: forearm pronation-supination and wrist flexion-extension. Each movement has three computer-controlled modes: (1) passive-passive, with both arms being moved by the machine with speed and range of motion individually adjustable; (2) active-passive, with the nonaffected arm driving the affected arm in a mirror-like fashion; and (3) active-active, with both arms actively moving against resistance. The speed of movement, the amount of resistance, and the range of movement can be adjusted individually. The device has a mechanical breaking of the movement when the torques exceeded 4 Nm, emergency breaks in the reach of the patients, skin friendly materials, and minimal risk for contusions.
  Other Names: Bi-Manu-Track; Reha-Stim Co., Berlin, Germany
  Arms: Robot-assisted therapy with Bi-Manu-Track (BMT)
Behavioral: Control intervention (CI) — he control group's therapy will be designed to control for the duration and intensity of the robot-assisted training (90 min/day, 5 days/wk, for 4 wk). The therapeutic activities in the control group will involve passive range of motion, weight bearing, stretching, strengthening of the paretic arm, gross motor activities, coordination tasks, unilateral and bilateral fine motor tasks, transition, mobility, and posture/balance.
  Arms: Control intervention group (CI)

SUMMARY:
Robot-assisted training (RT) devices developed to date have a significant impact on stroke rehabilitation. Several research groups have developed the robotic devices and examined their efficacy on improving UL function after stroke. All these robotic devices have been applied in stroke rehabilitation and their efficacy are evaluated, but the scientific evidence for the mechanisms of RT-induced recovery, the relative treatment effects of unilateral vs bilateral robotic trainings, and the impact on physiological responses is still lacking.

The primary purposes of this study are to examine (1) the relative immediate treatment effects of unilateral vs bilateral RT on motor impairments/performance and daily functions in patients with subacute stroke; (2) the long-term benefits of unilateral vs bilateral RT by conducting a 6-month follow up evaluation; and (3) the effects of RT on movement reorganization as well as on the physiological markers of inflammation, oxidative stress, erythrocyte deformability, and blood glucose. These overall findings will help better understanding of the efficacy of RT on functional outcomes, movement reorganization, and physiological markers. The investigators would additionally explore the possible differential treatment effects in patients with different levels of motor severity (i.e., moderate vs. severe).

The investigators hypothesize that (1) both unilateral (the InMotion3) and bilateral (the Bi-Manu-Track) robot-assisted training would bring larger benefits on motor performance and daily function than the control treatment; (2) such benefits would retain during the follow-up; (3) there would be differential immediate and retention effects of unilateral (the InMotion3) and bilateral (the Bi-Manu-Track) robot-assisted training on different outcome measures; (4) better movement reorganization as well as physiological marker expressions would be found in both robotic groups compared to control group; and (5) there would be differential effects of robotic therapy between participants with moderate vs. severe motor impairment.

DETAILED DESCRIPTION:
Subacute stroke participants will be recruited from the Chang Gung Memorial Hospital and then were randomly assigned to 1 of the 3 groups: RT with the InMotion3 (unilateral) robot group, RT with the Bi-Manu-Track (bilateral) robot group, and conventional intervention group.

Assessments on motor impairments/performance (Fugl Mayer Assessment, Modified Ashworth Scale, MyotonePRO, Medical Research Council scale, Jamar dynamometer, and Action Research Arm Test) and daily functions (Motor Activity Log, ABILHAND Questionnaire, accelerometer, and Adelaide Activities Profile) take about 40 minutes to complete. Kinematic evaluation will take about 1 hour. Blood samples of the patients (12 ml.) will be collected to examine the physiological markers (ie, inflammation-related markers, oxidative stress markers, erythrocyte deformability, and blood glucose) before and after intervention. A total of 24 ml blood will be collected in this study. Except for the blood taking, all the examinations are non-invasive.

Analysis of covariance (ANCOVA), controlling for the pretest differences, will be separately performed for each outcome measure to test the effects of different intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* first episode of stroke in cortical regions
* time since stroke less than 6 months and more than 2 weeks, i.e., subacute stage
* initial motor part of UE of FMA score ranging from 24 to 52, indicating moderate to severe movement impairment
* no serious cognitive impairment (i.e., Mini Mental State Exam score > 24)

Exclusion Criteria:

* aphasia that might interfere with understanding instructions
* chronic inflammatory, autoimmune and hematological disorders
* intake of anti-inflammatory drugs
* major health problems or poor physical conditions that might limit participation
* current participation in any other research

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Change of Kinematic analysis | Change from baseline in kinematic analysis immediately after the completion of intervention
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.
Changes of Fugl-Meyer Assessment (FMA) | Change from baseline in Fugl-Meyer Assessment immediately after the completion of intervention and at a 6-month follow-up
  The UE part of FMA will be used to evaluate sensorimotor impairment (Fugl Meyer et al., 1975). The motor part consists of 33 items for the reflexes and movement of shoulder, elbow, forearm, wrist, hand, and coordination/speed. Each item is scored on a scale of 0-2 with a maximum of 66 for the motor part. Higher score indicates a better reduction of motor impairment of UE. Satisfactory psychometric characteristics of FMA have been demonstrated (Hsueh & Hsieh, 2002; Platz et al., 2005).
Changes of Modified Ashworth Scale (MAS) | Changes from baseline in Modified Ashworth Scale immediately after the completion of intervention and at a 6-month follow-up
  The MAS is the most frequently used clinical rating scale to measure muscle spasticity. This measure involves manually moving a limb through the range of motion (ROM) to passively stretch specific muscle groups. The grades of spasticity in MAS are as follows: 0 = No increase in muscle tone; 1 = Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is(are) moved in flexion or extension; 1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2 = More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved; 3 = Considerable increase in muscle tone, passive movement difficult; 4 = Affected part(s) rigid in flexion or extension (Bohann & Smith, 1987).
Changes of MyotonPRO | Changes from baseline in MyotonPRO immediately after the completion of intervention and at a 6-month follow-up
  The Myoton is a hand-held device measure of three mechanical properties of muscle: tone, stiffness and elasticity (Viir et al., 2007). In this study, MyotonPRO will be mainly used to assess muscle tone of the arm. Muscle tone is characterized by the parameter in the Myoton: F - Frequency, Hz. The basic principle is the same in all prototypes but the MyotonPRO has several updates such as a triaxial accelerometer. MyotonPRO is more feasible than the earlier prototypes for application (Korhonen, Vain, Vanninen, Viir, & Jurvelin, 2005; Vain & Kums, 2002).
Changes of Medical Research Council scale (MRC) | Changes from baseline in Medical Research Council scale immediately after the completion of intervention and at a 6-month follow-up
  The muscle power of the affected arm will be examined by the MRC scale (Medical Research Council, 1976). The MRC Scale is reliable measurement with score ranged from 0 (no contraction) to 5 (normal power) (Gregson et al., 2000). The muscle strength of shoulder flexors/abductors, elbow flexors/extensors, wrist flexors/extensors, and finger extensors will be graded by the scale in this study.
Changes of the Jamar dynamometer | Changes from baseline in the Jamar dynamometer immediately after the completion of intervention and at a 6-month follow-up.
  The Jamar dynamometer is a standard, accurate, adjustable-handle tool specifically for measuring grip strength (Mathiowetz, Weber, Volland, & Kashman, 1984). Patients will sit with their shoulder adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral position, and wrist between 0° and 30° dorsiflexion and between 0° and 15° ulnar deviation. Patients will be asked to perform tasks under the unilateral and bilateral conditions. In the unilateral condition, patients will be asked to exert only with one hand (affected or "unaffected"); in the bilateral condition, patients will be asked to exert with both hands. Three trials will be taken at each assessment, and the average of three trials will be documented.
Changes of Action Research Arm Test (ARAT) | Changes from baseline in Action Research Arm Test immediately after the completion of intervention and at a 6-month follow-up
  ARAT will be used to assess the motor function of UE. A total of 19 items are to test the movement of grasp, grip, pinch, and gross motor, with a scale of 0-3 for each item (maximal of 57). Higher score refers to better motor function of UE. The ARAT has been found to have good psychometric properties (Hsueh & Hsieh, 2002).
Changes of Motor Activity Log (MAL) | Changes from baseline in Motor Activity Log immediately after the completion of intervention and at a 6-month follow-up
  MAL will be used to capture the level of use of affected UE in daily living. The MAL is a semi-structured interview assessing the amount of use (AOU) and quality of movement (QOM) of the affected arm in 30 main daily activities. It scores 0-5 for each activity. Higher score means better performance of affected arm. Study has demonstrated that MAL is an instrument with good internal consistency, interrater reliability, and construct validity (Uswatte et al., 2006).
Changes of ABILHAND Questionnaire | Changes from baseline in ABILHAND Questionnaire immediately after the completion of intervention and at a 6-month follow-up
  The ABILHAND Questionnaire will be used to evaluate the ability of UE in functional activities. There are 23 bimanual activities to measure subjectively perceived difficulty in performing some common activities in daily living, such as buttoning, cutting nails, and opening a bottle (Penta, Tesio, Arnould, Zancan, & Thonnard, 2001). It scores on a scale of 0-3 (0-cannot perform, 1-performs partially or with great difficulty, 2-performs with some difficulty, 3-performs fully). Its reliability and construct validity has been confirmed (Penta et al., 2001).
Change of Accelerometers | Change from baseline in accelerometers immediately after the completion of intervention
  This measure, quantitatively recording the amount of activity in free-living conditions, will be used to reflect the change in the amount of affected arm use over time. The participants will be asked to wear an accelerometer on each arm for 3 consecutive days to measure what they actually do before and immediately after treatment. In this project, acceleration will be sampled at 10 Hz and summed over a user-specified epoch. The recording epoch in this study will be 2 seconds; recording capacity will be approximately 72 hours. A "threshold-filter" will be applied to the raw recordings to obtain an accurate measure of the duration of arm movement. The ratio of the duration of the affected to the non-affected arm movement, used in this study, is a reliable and valid real-world measure of upper limb treatment outcome (Uswatte et al., 2006).
Changes of Adelaide Activities Profile (AAP) | Changes from baseline in Adelaide Activities Profile immediately after the completion of intervention and at a 6-month follow-up
  AAP will be applied to indicate the level of participation in household and community activities. This profile includes 21 activities in the four areas: domestic chores, household maintenance, service to others, and social activities. It scores on a scale of 0-3, with higher point meaning more frequent participation. The AAP is found to have good validity and reliability (Bond & Clark, 1998).

SECONDARY OUTCOMES:
Change of inflammatory markers | Change from baseline in inflammatory markers immediately after the completion of intervention
  Proinflammatory markers and anti-inflammatory markers will be used to reflect the changes on inflammation. Proinflammatory markers include C-reactive protein, tumor necrosis factor-α (TNF-α), interleukin (IL)-1β, IL-6, soluble intercellular adhesion molecule (sICAM), and matrix metalloproteinase 9 (MMP 9). Anti-inflammatory markers include IL-10 and IL-1 receptor antagonist.
Change of oxidative stress markers | Change from baseline in oxidative stress markers immediately after the completion of intervention
  Oxidative stress markers and antioxidative markers will be used to reflect the changes on oxidative stress. Oxidative stress makers include malondialdehyde (MDA), 8-Hydroxy-2-deoxyguanosine (8-OHdG), and immunoglobulin G (IgG), whereas antioxidants include superoxide dismutase (SOD), glutathione peroxidase (GPx), and catalase.
Change of erythrocyte deformability | Change from baseline in erythrocyte deformability immediately after the completion of intervention
  The Elongation Index (EI) will be used to determine the RBC deformability, which is based on an isointensity curve in the diffraction pattern by using an ellipse-fitting program. EI is calculated by (L-W)/(L+W), where L and W are the major and minor axes of the ellipse, respectively. The deformability index (δ) is defined as the ratio of the major to the minor axis length (L/W) (Shin, Ku, Park, & Suh, 2005).
Change of blood glucose indicators | Change from baseline in blood glucose indicators immediately after the completion of intervention
  Recent research indicates that the blood glucose levels of patients were significantly associated with stroke severity and functional outcomes after stroke (Hu et al., 2012; Martin, Ratan, Reding, & Olsen, 2012; Wu et al., 2012). To investigate the relationships between blood glucose levels and functional outcomes, we will also test the level of glucose and HbA1C for the participants before and after rehabilitation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kwei-Shan, Tao-Yuan, Taiwan